CLINICAL TRIAL: NCT01533233
Title: Safety and Results of Thoracoscopic Lobectomy Using Nonintubated Anesthesia Versus Intubated General Anesthesia for Lung Cancer Patients.
Brief Title: Thoracoscopic Lobectomy Using Nonintubated Anesthesia Versus Intubated General Anesthesia for Lung Cancer Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200911022R
Record Dates: First submitted 2011-02-15; First posted 2012-02-15 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Lung Cancer
Keywords: thoracoscopy; lung cancer; lobectomy; epidural anesthesia
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- nonintubated anesthesia (Experimental): Thoracoscopic lobectomy using nonintubated anesthesia
  Interventions: Procedure: thoracoscopic lobectomy and mediastinal lymph node dissection
- intubated general anesthesia (Active Comparator): Thoracoscopic lobectomy using intubated general anesthesia
  Interventions: Procedure: thoracoscopic lobectomy and mediastinal lymph node dissection

INTERVENTIONS:
Procedure: thoracoscopic lobectomy and mediastinal lymph node dissection
  Other Names: VATS lobectomy

SUMMARY:
The purpose of this study is to study the safety and results of thoracoscopic lobectomy using non-intubated thoracic epidural anesthesia versus intubated general anesthesia for lung cancer patients.

DETAILED DESCRIPTION:
Lung cancer is the leading cause of cancer death in Taiwan. Traditionally, open thoracotomy has been the standard approach for lung cancer surgery, including lobectomy and pneumonectomy. With the advance of thoracoscopic technique, thoracoscopic lobectomy has emerged as a reasonable option for the management of early-stage non-small cell lung cancer (NSCLC), and is supported by evidence-based treatment guidelines. Advantages of thoracoscopic lobectomy compared with thoracotomy include less postoperative pain, shorter hospitalization, and decreased postoperative pulmonary complications.

Traditionally, general anesthesia (GA) with one-lung ventilation using double-lumen endotracheal intubation has been considered mandatory in both open and thoracoscopic surgery. However, adverse effects of GA may occur after the operation, including ventilator-induced lung injury, impaired cardiac performance, postoperative nausea and vomiting, and residual neuromuscular blockade.

In order to reduce the adverse effects of GA, nonintubated anesthesia has been recently employed to perform thoracic surgery procedures including coronary artery bypass, management of pneumothorax, resection of pulmonary nodules and solitary metastases, lung volume reduction (LVR), and even transsternal thymectomy. The results achieved in these early series have been encouraging. In Taiwan, nonintubated thoracic surgery has also been performed at Taipei Veteran General Hospital in a high risk patient with satisfactory results.

The role of nonintubated anesthesia in thoracoscopic lobectomy is rarely investigated. There is a report showed that lobectomy using nonintubated anesthesia is safe and feasible, although only 3 cases were reported [13]. In our hospital, we also performed 6 thoracoscopic lobectomy using nonintubated anesthesia between August and October, 2009 with satisfactory results. Until now, the safety and effects of nonintubated anesthesia in thoracoscopic lobectomy has been unclear and comparison between nonintubated and intubated general anesthesia has never been reported. We hypothesize that nonintubated thoracoscopic lobectomy will be associated with a comparable oncological results, lower cardiopulmonary complications, and shorter intensive care unit (ICU) and hospital stays. To this end, we will compare safety and results of thoracoscopic lobectomy using nonintubated anesthesia versus intubated general anesthesia for lung cancer patients.

This study will be performed at National Taiwan University Hospital. A total of 100 patients will be included (50 patients in each arm).

ELIGIBILITY:
Inclusion Criteria:

1. Non-small cell lung cancer with clinical staging of I or II for whom thoracoscopic lobectomy is feasible.
2. Age between 25 and 80 years old
3. Tumor size < 5 cm without chest wall, diaphragm, or main bronchus invasion
4. Predicted FEV 1.0 > 60% or FEV1.0 > 1.5L
5. Organ Function Requirements:

   * Adequate hematological function (ANC > 1.5 x 109/L, platelets > 100 x 109/L)
   * PT, PTT<1.5X
6. Written inform consent

Exclusion Criteria:

1. Failed thoracic epidural catheter insertion
2. A history of previous epidural catheter insertion or ipsilateral thoracic operation
3. Signs of intrapleural adhesions
4. Pregnant or lactation female
5. ASA score greater than 3
6. Unfavorable airway or spinal anatomy judged by anesthesiologist
7. Sleep apnea

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Comparing the safety after intervention of each group. | 1 month
  Comparing the complication and morbidity after intervention of each group

SECONDARY OUTCOMES:
Short-term outcome | one month
  including ICU stay, period of ventilator use, hospital stay, number of days with chest drainage, adverse events, etc.
Oncological outcome | 5 years
  Number of LN dissection and overall survival after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Shing Chen, MD, PhD, Study Chair — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan